CLINICAL TRIAL: NCT01815580
Title: HIV Testing and Treatment to Prevent Onward HIV Transmission Among MSM and Transgender Women in Lima, Peru
Brief Title: HIV Test and Treat to Prevent HIV Transmission Among MSM and Transgender Women
Acronym: SABES?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Asociación Civil Impacta Salud y Educación, Peru (Other); Asociación Civil Via Libre, Peru (Other); Epicentro, Peru (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ann C Duerr, Professor (Member), Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TNT-Peru; R01DA032106 (NIH)
Record Dates: First submitted 2013-03-15; First posted 2013-03-21 (Estimated); Results first posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: HIV
Keywords: HIV; Treatment as Prevention; Seek, Test, Treat, Retain Strategies
MeSH Terms: interventions — Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate ART (Atripla or Stribild) (Active Comparator): Daily Atripla or Stribild will be provided to these patients for the duration of the study beginning at enrollment.
  Interventions: Drug: Atripla or Stribild
- Deferred ART (Atripla or Stribild) (Placebo Comparator): Daily Atripla or Stribild will be provided to these patients for the duration of the study beginning at 24 weeks.
  Interventions: Drug: Atripla or Stribild

INTERVENTIONS:
Drug: Atripla or Stribild — Antiretroviral therapy
  Other Names: (alternate: Truvada + 3rd ARV)

SUMMARY:
This study will recruit men and transgender women with acute or recent HIV infection. It wil look at how HIV medicines (ART) when given very early after HIV infection affect the amount of HIV in the blood, semen and rectal secretions. In addition, Investigators will be using modeling studies to look at whether or not this kind of HIV treatment can decrease the risk that a man will infect a person he has sex with and to find out how failure to take medications will impact spreading the virus to other people.

In this study, one group will be randomized (like a coin toss) to start ART immediately (just at the time of the enrollment visit) and the other group will wait until week 24 of the study to start ART. Both groups will be followed for a total of 48 weeks and will continue to receive ART from local sources after the study is over.

DETAILED DESCRIPTION:
This is three-step study. Step 1 will screen men who have sex with men (MSM) and transgender women who are unaware of their HIV status and 1) report high risk behaviors for acquiring HIV-1 infection or 2) who have symptoms of acute retroviral syndrome or 3) who have a sexual partner with newly-diagnosed acute or recent HIV infection. HIV testing will be conducted for several thousand MSM and transgender women from study opening until July 2015. In Step 2, high risk HIV-1 uninfected MSM and transgender women with high risk for acquiring HIV will be tested at regular intervals for incident HIV-1 (using tests for HIV p24 and/or HIV RNA). (During this period, men will receive standard HIV prevention interventions.) In Step 3, individuals with acute or recent HIV-1 infection will be enrolled in a 48-week randomized, open-label study of the effects of immediate vs. deferred ART on the decay dynamics of HIV viral load in plasma, semen and rectal secretions. (ART will be provided prior to 24 weeks for any participant in the deferred ART arm who meets initiation criteria.) All participants will be followed for 48 weeks after which they will continue ART from other sources.

ELIGIBILITY:
Inclusion Criteria:

* Adult men who have sex with men, and transgender women
* Unaware of HIV status at enrollment in follow-up cohort
* High risk for HIV infection
* Willing to test for HIV
* No prior ART, including prior administration of pre- and post-exposure prophylaxis in the last 30 days
* Willing to provide informed consent

Exclusion Criteria:

* Prior receipt of investigational anti-HIV vaccine
* Ongoing therapy with any of the following:

  1. Systemic corticosteroids. Short course less than or equal to 21 days of corticosteroids is allowed
  2. Systemic chemotherapeutic agents
  3. Nephrotoxic systemic agents, including aminoglycosides, amphotericin B, cidofovir, cisplatin, foscarnet, pentamidine
  4. Immunomodulatory treatments including Interleukin-2
  5. Investigational agents
* Known allergy/sensitivity or any hypersensitivity to components of study drugs (ART) or their formulations
* Active drug or alcohol use or dependence that would interfere with adherence to study requirements
* Serious medical or psychiatric illness that would interfere with the ability to adhere to study requirements
* Chronic or acute hepatitis B infection
* Use of female hormonal products based on estrogen or derivatives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Duerr, M.D., Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Asociación Civil Impacta Salud y Educación, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bachman VF, Montano MA, Ulrich A, Villaran M, Cabello R, Gonzalez P, Sanchez H, Lama JR, Duerr A. Correlates of condomless anal intercourse with different types of sexual partners among men who have sex with men and transgender women in Lima, Peru. AIDS Care. 2023 Jun;35(6):791-799. doi: 10.1080/09540121.2021.1994517. Epub 2021 Oct 26. PMID 34702087
- [Derived] Mayer ME, White E, Montano MA, Lama JR, Sanchez H, Cabello R, Sanchez J, Pasalar S, Duerr A. Sexual Behavior Among Men Who Have Sex With Men: The Need for More Targeted Outreach to Men Who Also Have Sex With Cisgender Women. J Acquir Immune Defic Syndr. 2021 Mar 1;86(3):265-270. doi: 10.1097/QAI.0000000000002568. PMID 33148993
- [Derived] Lama JR, Ignacio RAB, Alfaro R, Rios J, Cartagena JG, Valdez R, Bain C, Barbaran KS, Villaran MV, Pilcher CD, Gonzales P, Sanchez J, Duerr A. Clinical and Immunologic Outcomes After Immediate or Deferred Antiretroviral Therapy Initiation During Primary Human Immunodeficiency Virus Infection: The Sabes Randomized Clinical Study. Clin Infect Dis. 2021 Mar 15;72(6):1042-1050. doi: 10.1093/cid/ciaa167. PMID 32107526

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate ART (Atripla or Stribild) | Deferred ART (Atripla or Stribild)
Started | 110 | 115
Completed | 98 | 100
Not Completed | 12 | 15
Not completed — Lost to Follow-up | 4 | 7
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Excluded from analysis | 5 | 4

BASELINE CHARACTERISTICS:
Population: 5 participants from the Immediate arm and 4 participants from the Deferred arm were excluded from the analyses because by the time they were enrolled they could no longer be considered Acute or Recent HIV infection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate ART (Atripla or Stribild) | Deferred ART (Atripla or Stribild) | Total
Number analyzed (Participants) | 105 | 111 | 216
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.9 (7.3) | 26.6 (6.7) | 27.2 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 105 | 111 | 216
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 105 | 111 | 216
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Peru | 105 | 111 | 216
Baseline Viral Load [Mean (Standard Deviation); unit: Log10(copies/mL)] — This is a measure of the amount of HIV virus in the blood at the time of enrollment (Baseline).
  Log10(copies/mL) | 5.84 (1.16) | 5.78 (0.96) | 5.81 (1.06)
Baseline CD4 [Mean (Standard Deviation); unit: CD4 T Cell count/mm^3] — This is a measure of CD4 white blood cells in the blood at the time of enrollment (Baseline). A lower CD4 could indicate a more compromised immune system. Population: 2 participants in the Immediate arm and 1 participant in the deferred arm are missing a baseline CD4.
  CD4 T Cell count/mm^3
    number analyzed (Participants) | 103 | 110 | 213
    (all) | 430.1 (207.6) | 432.3 (212.3) | 431.2 (209.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HIV Viral Load Suppression in Plasma
Description: To quantify HIV viral load suppression (<1000 copies/mL) in plasma at Baseline and weeks 12, 24, 36, and 48 weeks Suppressed at Baseline = HIV Viral load measured at the time of enrollment was <1000 copies/mL Suppressed at Week 12 = HIV Viral load measured 12 weeks after enrollment was <1000 copies/mL etc.
Time Frame: Baseline, Week 12, Week 24, Week 36, and Week 48
Population: Not all participants had their viral load measured at all time points due to a missed visit or being lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate ART (Atripla or Stribild) | Deferred ART (Atripla or Stribild)
Number analyzed (Participants) | 105 | 111
Participants
  Suppressed at Baseline | 2 | 1
  Suppressed at week 12: number analyzed (Participants) | 98 | 104
  Suppressed at week 12 | 84 | 8
  Suppressed at week 24: number analyzed (Participants) | 95 | 104
  Suppressed at week 24 | 93 | 18
  Suppressed at week 36: number analyzed (Participants) | 96 | 99
  Suppressed at week 36 | 91 | 89
  Suppressed at week 48: number analyzed (Participants) | 95 | 98
  Suppressed at week 48 | 94 | 92

2. Primary Outcome: Number of Participants With HIV Viral Load Suppression in Semen
Description: To quantify HIV viral load suppression (<1000 copies/mL) in semen at Baseline and weeks 12, and, 24 weeks
Time Frame: Baseline, Week 12, and Week 24
Population: Analysis population is limited to study participants who gave both semen and plasma specimens. This was a planned subset of all participants. Not all participants had their semen viral load measured at all time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate ART (Atripla or Stribild) | Deferred ART (Atripla or Stribild)
Number analyzed (Participants) | 27 | 41
Participants
  Suppressed Baseline: number analyzed (Participants) | 19 | 33
  Suppressed Baseline | 4 | 7
  Suppressed week 12: number analyzed (Participants) | 24 | 31
  Suppressed week 12 | 21 | 17
  Suppressed week 24: number analyzed (Participants) | 20 | 23
  Suppressed week 24 | 19 | 9

3. Secondary Outcome: Sequence Clusters Identified Using Phylogenetic Analysis Among Participants With Early HIV Infection
Description: HIV present in blood samples from recently infected study participants was sequenced. Sequences that were similar to each other were grouped together in clusters. For this analysis, clusters were defined using a patristic distance threshold of 0.01, and a minimum cluster size of two.
Time Frame: HIV diagnosis visit
Measure: Count of Participants; unit: Participants
Groups:
- Not in Cluster: Clustering of HIV sequences used patristic-distance clustering (based on the sum of the branch lengths from one tip of the phylogenetic tree to another tip in the tree). ~700 nucleotides of the pol (partial reverse-transcriptase and partial protease) gene were used to construct phylogenetic trees. Participants in this group had pol gene sequences that were not within the conservative patristic distance threshold (0.01) of each other; a minimum cluster size of two was used.
- In a Cluster: Clustering of HIV sequences used patristic-distance clustering (based on the sum of the branch lengths from one tip of the phylogenetic tree to another tip in the tree). ~700 nucleotides of the pol (partial reverse-transcriptase and partial protease) gene were used to construct phylogenetic trees. Participants in this group had pol gene sequences that were within the conservative patristic distance threshold (0.01) of each other; a minimum cluster size of two was used.
Arm/Group | Not in Cluster | In a Cluster
Number analyzed (Participants) | 139 | 62
Participants
  Heavy drinker: Yes | 30 | 14
  Heavy drinker: No | 57 | 26
  Heavy drinker: Missing data | 52 | 22
  Audit Score >=20: Yes | 16 | 4
  Audit Score >=20: No | 117 | 49
  Audit Score >=20: Missing data | 6 | 9
  Any illicit drug use: Yes | 13 | 4
  Any illicit drug use: No | 126 | 58
  Any illicit drug use: Missing data | 0 | 0
  Sex Work: Yes | 16 | 5
  Sex Work: No | 123 | 56
  Sex Work: Missing data | 0 | 1
  Met a sex partner at any venue: Yes | 62 | 37
  Met a sex partner at any venue: No | 77 | 25
  Met a sex partner at any venue: Missing data | 0 | 0

4. Secondary Outcome: Percent of Participants Whose HIV Sequences Appear in Phylogenetically Defined Clusters
Description: as for outcome 3
Time Frame: HIV diagnosis visit
Population: Analysis population is limited to HIV-infected participants for whom HIV sequence data are available. Per initial protocol design, this analysis was conducted on all HIV sequences without dividing by randomization arm.
Measure: Number; unit: percentage of participants
Groups:
- Cluster Membership: Participants HIV sequenced
Arm/Group | Cluster Membership
Number analyzed (Participants) | 201
percentage of participants | 27

5. Secondary Outcome: Number of Participants Diagnosed With Acute HIV Infection Who Were Linked to Care
Description: To determine the proportion of individuals with evidence of acute infection (HIV-1 RNA-positive) who are successfully contacted for confirmatory HIV testing and are then linked to care.
Time Frame: within 3 months of diagnosis of acute HIV infection
Population: Analysis population includes only those participants whose HIV infection was diagnosed during the acute phase, that is prior to HIV seroconversion.
Measure: Count of Participants; unit: Participants
Groups:
- Acute: Participants with evidence of Acute HIV Infection
Arm/Group | Acute
Number analyzed (Participants) | 87
Participants | 71

6. Secondary Outcome: Partner Tracing
Description: Partner tracing and notification
Time Frame: within 3 months of diagnosis
Population: We were unable to trace potential partners because participants were unwilling or unable to identify recent partners
Measure: Count of Participants; unit: Participants
Groups:
- HIV Positive Participants: Participants with evidence of HIV Infection
Arm/Group | HIV Positive Participants
Number analyzed (Participants) | 216
Participants | 0

7. Secondary Outcome: Number of Participants Retained in Care
Description: To determine the number of participants who were retained in care at weeks 12, 24, 36, and 48
Time Frame: Baseline, Week 12, Week 24, Week 36, and Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate ART (Atripla or Stribild) | Deferred ART (Atripla or Stribild)
Number analyzed (Participants) | 105 | 111
Participants
  Retained at Week 12 | 102 | 106
  Retained at Week 24 | 101 | 105
  Retained at Week 36 | 98 | 103
  Retained at Week 48 | 96 | 101
Statistical Analysis 1: Comparison: Immediate ART (Atripla or Stribild) vs Deferred ART (Atripla or Stribild); Test type: Other; p > 0.75, Chi-squared

8. Secondary Outcome: Adherence to ART Regimen (Percentage of Pills Taken)
Description: To determine percentage of ART pills taken by participants randomized to immediate and deferred ART initiation.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: Percent of dispensed pills taken
Arm/Group | Immediate ART (Atripla or Stribild) | Deferred ART (Atripla or Stribild)
Number analyzed (Participants) | 105 | 111
Percent of dispensed pills taken | 93.6 (4.7) | 91.5 (13.4)
Statistical Analysis 1: Comparison: Immediate ART (Atripla or Stribild) vs Deferred ART (Atripla or Stribild); Test type: Other; p = 0.14, t-test, 2 sided

9. Secondary Outcome: Adherence to Viral Load (VL) Procedure
Description: To determine the number of participants who had a viral load test at Baseline and weeks 12, 24, 36, and 48
Time Frame: Baseline, Week 12, Week 24, Week 36, and Week 48
Population: Participants still in follow up at each time point who provided viral load measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate ART (Atripla or Stribild) | Deferred ART (Atripla or Stribild)
Number analyzed (Participants) | 105 | 111
Participants
  VL at Baseline | 105 | 111
  VL at Week 12: number analyzed (Participants) | 100 | 109
  VL at Week 12 | 98 | 104
  VL at Week 24: number analyzed (Participants) | 100 | 107
  VL at Week 24 | 95 | 104
  VL at week 36: number analyzed (Participants) | 99 | 103
  VL at week 36 | 96 | 99
  VL at Week 48: number analyzed (Participants) | 98 | 100
  VL at Week 48 | 95 | 98
Statistical Analysis 1: Comparison: Immediate ART (Atripla or Stribild) vs Deferred ART (Atripla or Stribild); Test type: Other; p > 0.3, Chi-squared

10. Secondary Outcome: Adherence to CD4 Procedure
Description: To determine the number of participants who had a CD4 test at Baseline and weeks 12, 24, 36, and 48
Time Frame: Baseline, Week 12, Week 24, Week 36, and Week 48
Population: Participants still in follow up at each time point who provided a CD4 measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate ART (Atripla or Stribild) | Deferred ART (Atripla or Stribild)
Number analyzed (Participants) | 105 | 111
Participants
  CD4 at Baseline | 103 | 110
  CD4 at Week 12: number analyzed (Participants) | 100 | 109
  CD4 at Week 12 | 99 | 104
  CD4 at Week 24: number analyzed (Participants) | 100 | 107
  CD4 at Week 24 | 97 | 104
  CD4 at Week 36: number analyzed (Participants) | 99 | 103
  CD4 at Week 36 | 97 | 100
  CD4 at Week 48: number analyzed (Participants) | 98 | 100
  CD4 at Week 48 | 96 | 98
Statistical Analysis 1: Comparison: Immediate ART (Atripla or Stribild) vs Deferred ART (Atripla or Stribild); Test type: Other; p > 0.12, Chi-squared

11. Secondary Outcome: Adherence to Questionnaires
Description: To determine the number of participants who completed the Computer Assisted Self interviews (CASI) at Baseline and weeks 12, 24, 36, and 48
Time Frame: Baseline, Week 12, Week 24, Week 36, and Week 48
Population: Participants still in follow up at each time point who completed the study questionnaires
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate ART (Atripla or Stribild) | Deferred ART (Atripla or Stribild)
Number analyzed (Participants) | 105 | 111
Participants
  CASI at Baseline | 100 | 109
  CASI at Week 12: number analyzed (Participants) | 100 | 109
  CASI at Week 12 | 96 | 102
  CASI at Week 24: number analyzed (Participants) | 100 | 107
  CASI at Week 24 | 95 | 100
  CASI at Week 36: number analyzed (Participants) | 99 | 103
  CASI at Week 36 | 92 | 99
  CASI at Week 48: number analyzed (Participants) | 98 | 100
  CASI at Week 48 | 90 | 92
Statistical Analysis 1: Comparison: Immediate ART (Atripla or Stribild) vs Deferred ART (Atripla or Stribild); Test type: Other; p > 0.22, Chi-squared

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Immediate ART (Atripla or Stribild) | Deferred ART (Atripla or Stribild)
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/111
Serious Adverse Events (participants affected / at risk) | 2/105 | 1/111
Other Adverse Events (participants affected / at risk) | 26/105 | 28/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate ART (Atripla or Stribild) (N=105) | Deferred ART (Atripla or Stribild) (N=111)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Suicidal attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate ART (Atripla or Stribild) (N=105) | Deferred ART (Atripla or Stribild) (N=111)
Proctitis chlamydial (Infections and infestations) | 8 (9) | 13 (16)
Proctitis gonococcal (Infections and infestations) | 10 (10) | 12 (13)
Syphilis (Infections and infestations) | 14 (16) | 13 (13)
Genitourinary chlamydia infection (Infections and infestations) | 4 (4) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 8 (9)
Genitourinary tract gonococcal infection (Infections and infestations) | 3 (3) | 6 (6)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8)
Proctitis (Gastrointestinal disorders) | 2 (2) | 6 (7)
Urethritis (Infections and infestations) | 3 (3) | 7 (8)
Hemorrhoids (General disorders) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT01815580/Prot_SAP_000.pdf